CLINICAL TRIAL: NCT01264081
Title: A Phase II Study of Lapatinib for the Treatment of Stage IV Melanoma Harboring ERBB4 Mutations
Brief Title: Lapatinib in Stage IV Melanoma With ERBB4 Mutations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol would not be able to reach stated accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Udo Rudloff, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110048; 11-C-0048
Record Dates: First submitted 2010-12-18; First posted 2010-12-21 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Malignant Melanoma
Keywords: Lapatinib; Melanoma; ERBB4 Mutation; Malignant Melanoma; Skin Cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lapatinib (Experimental): Lapatinib will be administered as an oral dose of 500 mg twice daily in the morning and evening one hour before or after meals.
  Interventions: Drug: Lapatinib

INTERVENTIONS:
Drug: Lapatinib — 500 mg PO (orally) twice a day for 28 days (1 cycle). Up to 27 cycles allowed if response seen.

SUMMARY:
Background:

- Studies of melanoma tumor samples have shown that tumor cells from approximately 20 percent of melanoma patients contain a specific mutation of a gene involved in making a protein called ERBB4, and that changes in this gene have been associated with cancer. Lapatinib, a drug that is currently approved for the treatment of breast cancer, has been shown in the laboratory to significantly slow the growth of melanoma cells that contain this specific ERBB4 gene mutation. Researchers are interested in determining whether lapatinib can be effective against melanoma in individuals who have the ERBB4 mutation.

Objectives:

- To evaluate the safety and effectiveness of lapatinib as a treatment for melanoma with ERBB4 mutation that has not responded to standard therapy.

Eligibility:

- Individuals at least 18 years of age who have stage 4 melanoma that has not responded to standard therapy.

Design:

* Participants will be screened with a full physical examination and medical history, as well as tests of tumor tissue taken from previous surgeries or biopsies or from a new biopsy that will be conducted before the start of the study. Test results to determine eligibility will be available within about 2 weeks.
* Participants will take four lapatinib tablets daily (two in the morning, 1 hour before or after breakfast and two in the evening, 1 hour before or after dinner) during every 28-day cycle of treatment. Participants will keep a medication diary to record tablets taken and any side effects from the medication.
* After the first 2 weeks, and every 2 to 4 weeks afterward for the first 12 weeks, participants will have clinic visits with blood samples and other tests to determine if lapatinib is causing their disease to shrink or be controlled. If the disease has not progressed, participants will continue to receive a new lapatinib supply every 28 days for up to 2 years (27 cycles), and will continue to have regular clinic visits to monitor the progress of treatment.
* When tumor tissue is easily accessible and can be easily biopsied, researchers will collect two additional biopsies, one after 2 weeks of treatment and one after 12 weeks of treatment....

DETAILED DESCRIPTION:
Background:

* Patients with stage IV melanoma have few available treatment options and an overall poor prognosis.
* Pre-clinical evidence suggests that lapatinib has activity against metastatic melanoma harboring ERBB4 mutations.

Objectives:

Primary Objectives:

-Determine the response rate to lapatinib administered as 500 mg orally twice daily on a continuous schedule in patients with metastatic melanoma harboring ERBB4 mutations.

Secondary Objectives:

* To determine the progression free survival of patients with stage IV melanoma treated with lapatinib monotherapy.
* To evaluate the safety of lapatinib in patients with metastatic melanoma
* To determine the impact of additional genetic alterations on the response to lapatinib in melanoma harboring ERBB4 mutations
* To develop a clinically applicable biomarker predictive of response to lapatinib in patients with melanoma harboring ERBB4 mutations
* To determine the pharmacokinetics of lapatinib administered as 500 mg orally twice daily on a continuous schedule in patients with metastatic melanoma harboring ERBB4 mutations

Eligibility:

* Patients greater than or equal to 18 years of age with stage IV melanoma, who have measurable disease and whose tumors express up to two ERBB4 gene mutations.
* Patient must be Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 1 and a life expectancy of more than 3 months.
* Patients must have adequate organ function.
* Patients must not have had surgery, chemotherapy, hormonal therapy, radiation therapy, or biological therapy for at least 4 weeks prior to starting study medication.
* Patients must not have an acute, critical illness.
* All patients who are sexually active and able to conceive will be required to use contraception during treatment with lapatinib.

Design:

* Patients will be screened for the presence of ERBB4 gene mutations in their tumor and only patients who harbor less than or equal to 2 ERBB4 mutations will be enrolled in the treatment phase of the study.
* Lapatinib will be administered as an oral dose of 500 mg twice daily (in the morning and evening) taken one hour before or after meals. Lapatinib will be given continuously; one cycle equals 28 days. Course 1 equals cycle 1; all subsequent courses are 8 weeks long (2 cycles). A patient may receive up to 27 cycles (14 courses).
* Up to 25 patients (allowing for a staged accrual of initially 16 patients who will receive lapatinib and are evaluable after the 1st cycle) will be enrolled over 2-3 years and the trial will be completed over 3-5 years, allowing for completion of follow-up.
* The primary objective of the trial will be to determine whether lapatinib monotherapy in this setting is able to be associated with a response rate (Partial Response (PR) + Complete Response (CR)) that can rule out 10% (p0=0.10) in favor of an improved response rate of 30% (p1=0.30).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed stage IV cutaneous melanoma.
* Patients must have measurable disease defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be greater than 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or greater than 20 mm when measured by chest x-ray. Lymph nodes must be greater than 15 mm in short axis when measured by CT or MRI.
* Patients must have no more than two oncogenic somatic ERBB4 mutations detected in one of the 28 exons of the ERBB4 gene analyzed from the tumor and which is not present in the matched normal deoxyribonucleic acid (DNA) as confirmed by sequence analysis of tumor genomic DNA derived from any biopsy specimen obtained at the participating clinical sites. Sequence analysis will be performed at the National Institutes of Health (NIH) Clinical Molecular Profiling Core, a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.

Note: Patients with 3 or more mutations in their ERBB4 gene may have an increased resistance to lapatinib and are not eligible for lapatinib treatment

* Patients must not have had chemotherapy, molecular therapy with B-RAF, mouse embryonic fibroblast (MEK), or c-kit inhibitors, hormonal therapy, radiation therapy, or biological therapy for at least 4 weeks prior to starting study medication. Patients who received mitomycin C, nitrosoureas, anti-cytotoxic T-lymphocyte antigen 4 (CTLA-4), or carboplatin must be 6 weeks from the last administration of therapy. Patients must have recovered from any acute toxicity related to prior therapy or surgery, to a grade 1 or less unless specified.
* Patients with no more than 3 intracranial metastases, which have been definitively treated by surgery or radiation therapy may be eligible for study provided there is no evidence of active disease for at least 2 months and no requirement for anticonvulsant therapy or steroids following treatment.
* Age greater than or equal to 18 years.

Note: Because no dosing or adverse event data are currently available on the use of lapatinib in patients less than 18 years of age, children are excluded from this study but will be eligible for future pediatric single-agent trials, if applicable.

* Life expectancy of greater than 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1 (Karnofsky greater than or equal to 70%).
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin within normal institutional limits
  * Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase (SGOT))/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase (SGPT)) less than or equal to 3 times institutional upper limit of normal
  * creatinine less than or equal to institutional upper limit of normal

OR

--creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.

* Patients must be willing to return to the Clinic for follow-up visits.
* Women of childbearing potential must have a negative beta-human chorionic gonadotropin (HCG) (serum or urine) within 14 days prior to study treatment and must be willing to practice effective birth control to prevent pregnancy while receiving treatment and for four months after treatment is discontinued. All males of child fathering potential must also be willing to practice effective birth control.

Note: Lapatinib is a tyrosine kinase inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lapatinib, breastfeeding should be discontinued if the mother is treated with lapatinib. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treating physician immediately.

* Ability to understand and the willingness to sign the Informed Consent Document.
* Patients who agree to participate in the pharmacokinetics (PK) portion of the study must be able to swallow lapatinib tablets for the duration of the PK studies.

EXCLUSION CRITERIA:

* Patients may not be currently receiving any other investigational agents.
* Patients may not have received prior treatment with tyrosine kinase inhibitors (e.g., lapatinib erlotinib, or gefitinib).
* Patients currently receiving any medication known to induce/inhibit cytochrome P450 3A4 (CYP3A4) as listed in Appendix D, which in the opinion of the principal investigator, would make the administration of study drug hazardous. Note: patients receiving any strong or moderate CYP3A4 inhibitors will be excluded.
* Patients with active hepatic or biliary disease (with exception of patients with Gilberts syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Human immunodeficiency virus (HIV)-positive patients on antiretroviral therapy are excluded because most antiretrovirals are strong or moderate CYP3A4 inhibitors.
* Any underlying medical condition which, in the opinion of the principal investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events
* Patients with any other concurrent malignancy, except for the following:

  * adequately treated basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix, or any other cancer from which the patient has been disease-free for five (5) years or more.

INCLUSION OF WOMEN AND MINORITIES:

Both men and women and members of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-05-20 (Actual); Primary Completion 2013-11-22 (Actual); Study Completion 2013-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Udo Rudloff, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies MA, Samuels Y. Analysis of the genome to personalize therapy for melanoma. Oncogene. 2010 Oct 14;29(41):5545-55. doi: 10.1038/onc.2010.323. Epub 2010 Aug 9. PMID 20697348
- [Background] Prickett TD, Agrawal NS, Wei X, Yates KE, Lin JC, Wunderlich JR, Cronin JC, Cruz P, Rosenberg SA, Samuels Y. Analysis of the tyrosine kinome in melanoma reveals recurrent mutations in ERBB4. Nat Genet. 2009 Oct;41(10):1127-32. doi: 10.1038/ng.438. Epub 2009 Aug 30. PMID 19718025
- [Background] Geyer CE, Forster J, Lindquist D, Chan S, Romieu CG, Pienkowski T, Jagiello-Gruszfeld A, Crown J, Chan A, Kaufman B, Skarlos D, Campone M, Davidson N, Berger M, Oliva C, Rubin SD, Stein S, Cameron D. Lapatinib plus capecitabine for HER2-positive advanced breast cancer. N Engl J Med. 2006 Dec 28;355(26):2733-43. doi: 10.1056/NEJMoa064320. PMID 17192538
- [Result] Kerkar SP, Kemp CD, Duffy A, Kammula US, Schrump DS, Kwong KF, Quezado M, Goldspiel BR, Venkatesan A, Berger A, Walker M, Toomey MA, Steinberg SM, Giaccone G, Rosenberg SA, Avital I. The GYMSSA trial: a prospective randomized trial comparing gastrectomy, metastasectomy plus systemic therapy versus systemic therapy alone. Trials. 2009 Dec 23;10:121. doi: 10.1186/1745-6215-10-121. PMID 20030854

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty participants were registered, tested for the ERBB4 mutation, and taken off study as screening failures as they did not have the ERBB4 mutation to be treated with Lapatinib.
Period: Participants Screened
Arm/Group | Lapatinib
Started | 34
Completed | 4
Not Completed | 30
Not completed — Screening failures | 30
Period: Started Treatment
Arm/Group | Lapatinib
Started | 4
Completed | 2
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Not complete cycle 1 due to death | 1
Period: Analysis
Arm/Group | Lapatinib
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lapatinib
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With a Partial Response (PR) and Complete Response (CR) to Lapatinib Who Have Metastatic Melanoma Harboring ERBB4 Mutations.
Description: The count of participants with a partial response and complete response is defined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The appearance of one or more new lesions is also considered progressions.
Time Frame: 3 years
Population: Only two participants could be evaluated for response and they had SD (none with a PR or CR). Other participants did not reach the evaluation point (i.e. discontinued Lapatinib)as per study protocol, therefore not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib
Number analyzed (Participants) | 2
Participants
  Partial Response | 0
  Complete Response | 0
  Stable Disease | 2
  Progressive Disease | 0

2. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately, 3 years
Population: Three study participants were affected by the adverse events: 2 - who completed the study and 1 who did not complete cycle 1 due to death of progressive disease. The participant who withdrew from study didn't take Lapatinib and experience any adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Lapatinib
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately, 3 years.
Description: Three study participants were affected by the adverse events: 2 - who completed the study and 1 who did not complete cycle 1 due to death of progressive disease. The participant who withdrew from study didn't take Lapatinib and experience any adverse events.
Arm/Group | Lapatinib
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib (N=3)
Thromboembolic event (Vascular disorders) | 1 (1) — Pulmonary embolus
Death NOS (General disorders) | 2 (2) — Death due to progressive disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lapatinib (N=3)
Rash maculo-paular (Skin and subcutaneous tissue disorders) | 2 (2) — Skin and subcutaneous tissue disorders
Agitation (Psychiatric disorders) | 1 (1) — Psychiatric disorders

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-02-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT01264081/Prot_SAP_000.pdf
  • Informed Consent Form (2012-02-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT01264081/ICF_001.pdf